CLINICAL TRIAL: NCT07101484
Title: A Study of GD007 (Human iPSC-Exosome Liquid Dressing) for Safety and Dose-Finding in Moderate-Severe Intrauterine Adhesion
Brief Title: A Study of GD007 (Human iPSC-Exosome Liquid Dressing) for Safety and Dose-Finding in Moderate-Severe Intrauterine Adhesions
Acronym: GD007
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT_ iPSC-Exosome Liquid Dress; 2024-SR-1162 (Other: Jiangsu Provincial People's Hospital EC Approval Number)
Record Dates: First submitted 2025-06-26; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: Moderate-Severe Intrauterine Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose drug group (Experimental): Low-dose Intervention Group for moderate-to-severe intrauterine adhesions
  * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Interventions: Drug: GD007 Low-dose drug group
- Mid-dose drug group (Experimental): * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Interventions: Drug: GD007 Mid-dose drug group
- High-dose drug group (Experimental): * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Interventions: Drug: GD007 High-dose drug group
- Blank Control drug group (Placebo Comparator): * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Interventions: Drug: GD007 Blank Control drug Group

INTERVENTIONS:
Drug: GD007 Low-dose drug group — o Eligible patients who provide informed consent will receive:
  * First exosome perfusion: 24 hours post-operatively
  * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Other Names: GD007
  Arms: Low-dose drug group
Drug: GD007 Mid-dose drug group — * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Other Names: GD007
  Arms: Mid-dose drug group
Drug: GD007 High-dose drug group — * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Other Names: GD007
  Arms: High-dose drug group
Drug: GD007 Blank Control drug Group — * Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.
  * Eligible patients who provide informed consent will receive:
    * First exosome perfusion: 24 hours post-operatively
    * Subsequent perfusions: Every 3 days (total 3 perfusions)
  Other Names: GD007
  Arms: Blank Control drug group

SUMMARY:
Intrauterine adhesions (IUA) remain highly prevalent in China, with incidence rates steadily increasing due to the rising number of intrauterine procedures. Literature reports indicate that IUA caused by repeated induced abortions, curettage, postpartum infections, and other intrauterine surgeries occurs in 25%-30% of cases, making it a leading cause of reduced menstrual flow, cyclic abdominal pain, recurrent miscarriage, and secondary infertility, significantly impairing women's reproductive health and overall well-being.

Currently, no effective treatment exists for severe IUA to fully restore fertility and normal menstrual physiology. The commonly used hysteroscopic adhesiolysis (TCRA) has a high recurrence rate of 62.5%, with a post-operative pregnancy success rate of only 22.5%-33.3%. Therefore, there is an urgent clinical need to explore novel therapeutic strategies for severe intrauterine adhesions.

Exosomes derived from induced pluripotent stem cells (iPS-Exo) offer significant advantages over MSC-derived exosomes due to their clonal origin, ensuring superior batch-to-batch consistency and stability. This feature enables more stringent quality control standards and facilitates standardized, scalable production and quality management systems. Compared to mesenchymal stem cells (MSCs) or MSC-derived exosomes, iPS-Exo exhibit multiple superior properties:

1. Higher potency of bioactive components:

   * As iPSCs represent an earlier differentiation stage than MSCs, iPS-Exo contain elevated levels of functional factors such as TGF-β (anti-inflammatory), BDNF (neurotrophic), and others.
   * Demonstrated biological effects:

     * Anti-apoptosis
     * Inflammation suppression
     * Angiogenesis promotion
     * Fibrosis inhibition
     * Enhanced tissue repair potential
2. Enhanced pharmaceutical suitability:

   * Clonal expansion ensures product homogeneity and manufacturing reproducibility.
   * Simplified quality control metrics compared to heterogeneous MSC-Exo.
3. Genetic engineering compatibility:

   o Amenable to precision modification for targeted therapeutic enhancement.
4. Preclinical efficacy evidence:

   * Neuroprotection: Superior to MSC-Exo in mitigating neuronal damage induced by oxygen-glucose deprivation and hydrogen peroxide-induced oxidative stress.
   * Epilepsy models: Significant reduction in seizure frequency/severity and decreased cerebral IL-6/TNF-α levels in treated mice.
   * Stroke models: Intravenous administration:

     * Suppressed Th1/Th17 immune responses post-ischemia
     * Increased Treg cell proportion
     * Modulated immune microenvironment
     * Reduced infarct volume and improved motor function
     * Enhanced survival rates Compared to small-molecule drugs or MSC-Exo with limited mechanisms, iPS-Exo demonstrate broader therapeutic potential for ischemic stroke, drug-resistant epilepsy, and other disorders. However, their application in treating endometrial damage from intrauterine adhesions (IUA) remains unexplored to date.

Goodain (Beijing) Pharmaceutical Technology Co., Ltd., a biotechnology company specializing in induced pluripotent stem cells (iPSCs) and exosome technologies, holds GMP laboratory certification. The company has independently developed clinical-grade iPSC-derived exosomes (iPS-Exo), which have been investigated in four investigator-initiated exploratory clinical trials across different indications, with no reported adverse events (AEs) or serious adverse events (SAEs) to date.

Preclinical Rationale

Our research team previously conducted preclinical studies using umbilical cord mesenchymal stem cell-derived exosomes (MSC-Exo) in a rat model of intrauterine adhesions (IUA). Results demonstrated that:

• Intrauterine perfusion of MSC-Exo significantly promoted:

* Endometrial regeneration in mechanically injured rats
* Increased endometrial gland density
* Enhanced cellular proliferation
* Higher embryo implantation rates These findings support the translational potential of exosome-based therapies for IUA.

Study Objective

Building on this preclinical evidence, we propose the first-in-human safety evaluation of clinical-grade iPS-Exo for moderate-to-severe IUA. This study aims to:

1. Establish preliminary safety profiles
2. Explore therapeutic efficacy signals
3. Address the unmet clinical need in severe IUA management Key Advantages

   * Regulatory-ready: GMP-certified production ensures batch consistency.
   * Clinical precedence: Favorable safety data from prior exploratory trials.
   * Mechanistic validation: Proven endometrial repair effects in animal models.

DETAILED DESCRIPTION:
1、Study Objectives

1. Primary Objective To evaluate the clinical safety of human iPSC-derived exosome liquid dressing (GD007) in patients with moderate-to-severe intrauterine adhesions (IUA).
2. Secondary Objectives To assess the IUA recurrence rate within 6 months post-treatment. To investigate endometrial thickness improvement as a marker of endometrial regeneration.

2、Study Design: Single-center, prospective, open-label 3、Study Procedures IUA Treatment Protocol Patients diagnosed with moderate-to-severe intrauterine adhesions (IUA) will undergo standard hysteroscopic adhesiolysis.

Eligible patients who provide informed consent will receive:

* First exosome perfusion: 24 hours post-operatively
* Subsequent perfusions: Every 3 days (total 3 perfusions)

Follow-up hysteroscopy at 1 month to assess adhesion recurrence:

If adhesions recur: Repeat adhesiolysis (Step 1) followed by another 3-perfusion cycle (24h post-op)

Monthly follow-up for 6 months to monitor:

* Adverse events (per CTCAE v5.0)
* Endometrial thickness (transvaginal ultrasound) Fertility Management IVF/ICSI:Embryo transfer performed per standard protocols after completing exosome therapy Endometrial preparation and transfer procedures follow institutional SOPs Natural conception:Ultrasound-guided ovulation monitoring + timed intercourse Detailed documentation of clinical pregnancy outcomes 4、 Patient Selection Criteria Inclusion Criteria 1) Demographics

  * Females aged 20-40 years with fertility desire 2) Diagnostic Confirmation
  * Hysteroscopically confirmed moderate-to-severe intrauterine adhesions (IUA) *(Per 2015 Chinese IUA Scoring System: Moderate=9-18 points; Severe=19-28 points)* 3) Surgical Eligibility
  * Indicated for hysteroscopic surgery without contraindications 4) Ovarian Function
  * Normal ovarian reserve (AMH ≥1.1 ng/mL or AFC ≥5) 5) Consent
  * Voluntary participation with signed informed consent Exclusion Criteria

    1. Active Infections
  * Acute pelvic inflammatory disease or vaginitis 2. Uterine Abnormalities
  * History of uterine artery embolization
  * Submucosal fibroids (>2 cm)
  * Adenomyosis with uterine size >8-week gestation 3. Neoplastic Conditions
  * Malignancies
  * Endometrial hyperplasia (with/without atypia) 4. Contraindications
  * Hypersensitivity to hyaluronic acid gel 5. Hormonal Medications
  * Chronic steroid use
  * High-dose hormone therapy (>8 mg/day estrogen/progestin within 1 month) 6. Hematologic Disorders
  * Thrombocytopenia (platelets <50×10⁹/L)
  * Coagulopathy (aPTT >1.5×ULN) 7. Systemic Diseases
  * Uncontrolled diabetes (HbA1c >7%)
  * Severe cardiovascular disease (NYHA Class III/IV)
  * Life-threatening comorbidities 8. Clinical Trial Participation
  * Enrollment in other interventional trials within 3 months
  * Recent drug trials (<5 half-lives from last dose) 9. Investigator's Discretion
  * Any condition deemed unsuitable for participation

ELIGIBILITY:
Inclusion Criteria:

* 1) Demographics

  * Females aged 20-40 years with fertility desire 2) Diagnostic Confirmation
  * Hysteroscopically confirmed moderate-to-severe intrauterine adhesions (IUA) *(Per 2015 Chinese IUA Scoring System: Moderate=9-18 points; Severe=19-28 points)* 3) Surgical Eligibility
  * Indicated for hysteroscopic surgery without contraindications 4) Ovarian Function
  * Normal ovarian reserve (AMH ≥1.1 ng/mL or AFC ≥5) 5) Consent
  * Voluntary participation with signed informed consent

Exclusion Criteria:

1. Active Infections

   o Acute pelvic inflammatory disease or vaginitis
2. Uterine Abnormalities

   * History of uterine artery embolization
   * Submucosal fibroids (>2 cm)
   * Adenomyosis with uterine size >8-week gestation
3. Neoplastic Conditions

   * Malignancies
   * Endometrial hyperplasia (with/without atypia)
4. Contraindications

   o Hypersensitivity to hyaluronic acid gel
5. Hormonal Medications

   * Chronic steroid use
   * High-dose hormone therapy (>8 mg/day estrogen/progestin within 1 month)
6. Hematologic Disorders

   * Thrombocytopenia (platelets <50×10⁹/L)
   * Coagulopathy (aPTT >1.5×ULN)
7. Systemic Diseases

   * Uncontrolled diabetes (HbA1c >7%)
   * Severe cardiovascular disease (NYHA Class III/IV)
   * Life-threatening comorbidities
8. Clinical Trial Participation

   * Enrollment in other interventional trials within 3 months
   * Recent drug trials (<5 half-lives from last dose)
9. Investigator's Discretion o Any condition deemed unsuitable for participation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Reproductive-aged women (20-40 years) desiring fertility
Enrollment: 29 (Estimated)
Dates: Start 2025-05-04 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Measure: Incidence of severe intolerability after intrauterine perfusion of iPS cell-derived exosome liquid dressing | From Day 1 of GD007 exosome dressing application to 6 months post-treatment
  including:
  * Persistent severe nausea/vomiting
  * Rash
  * Fever
  * Acute reproductive tract infections
  * Severe abnormal uterine bleeding (non-surgical etiology)

SECONDARY OUTCOMES:
Effectiveness measures: Recurrence rate of intrauterine adhesions (IUA) post-treatment | From Day 1 of GD007 exosome dressing application to 6 months post-treatment
  Recurrence rate of intrauterine adhesions (IUA) post-treatment: The rate of IUA recurrence detected by hysteroscopy after the first treatment with iPS cell-derived exosome liquid dressing following initial adhesiolysis.
Effectiveness measures:Endometrial thickness | From Day 1 of GD007 exosome dressing application to 6 months post-treatment
  Endometrial thickness: Change in endometrial thickness (measured by ultrasound on the day of HCG transformation) before and after intrauterine perfusion of iPS cell-derived exosomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Center o Reproductive Medicine of First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Share Study Protocol Approved by the Institutional Ethics Committee and Final Clinical Study Report with Investigator Signatures
Supporting Information: Study Protocol